CLINICAL TRIAL: NCT00879190
Title: Comparison of Ampicillin / Sulbactam vs. Ampicillin / Gentamicin for Treatment of Intrapartum Chorioamnionitis: a Randomized Controlled Trial
Brief Title: Ampicillin / Sulbactam vs. Ampicillin / Gentamicin for Treatment of Chorioamnionitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natali Aziz, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-03192009-2018; 15562 (Other: Stanford University Research Compliance Office)
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Chorioamnionitis
MeSH Terms: conditions — Chorioamnionitis | interventions — sultamicillin; Ampicillin; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unasyn (ampicillin/sulbactam) (Active Comparator)
  Interventions: Drug: Unasyn
- Ampicillin/gentamicin (Active Comparator)
  Interventions: Drug: Ampicillin/gentamicin

INTERVENTIONS:
Drug: Unasyn — Unasyn 3 grams intravenously every 6 hours, plus intravenous normal saline placebo dose every 8 hours until 24 hours post delivery.
  Arms: Unasyn (ampicillin/sulbactam)
Drug: Ampicillin/gentamicin — Gentamicin 1.5mg/kg intravenously every 8 hours plus ampicillin 2 grams intravenously every 6 hours until 24 hours post delivery.
  Arms: Ampicillin/gentamicin

SUMMARY:
Chorioamnionitis is an infection of the placenta and amniotic membranes (bag of waters) surrounding the baby inside of a pregnant woman prior to delivery. This infection is somewhat common and is routinely treated with antibiotics given to the mother both before and after the baby is born. Currently it is not known what is the best choice of antibiotics to treat this type of infection, but commonly used treatments include Unasyn (ampicillin/sulbactam) or ampicillin/gentamicin. We plan to compare these two different antibiotic regimens to see if one is better than the other at treating and preventing bad outcomes from chorioamnionitis in women and babies.

DETAILED DESCRIPTION:
Patients who meet inclusion criteria will be approached upon admission to Labor and Delivery. A study staff member will describe the study and offer participation. If a patient agrees to participate, she will sign research protocol and HIPAA consent forms and receive a copy of these forms. The patient's chart will be flagged, indicating that she is a study participant. The patient's prenatal care and labor and delivery will be managed by her physician per standard of care at the physician's discretion, including routine intrapartum treatment of Group B streptococcus (GBS) colonization using ampicillin. When a participating patient is diagnosed with chorioamnionitis, she will be randomized in a blinded fashion to Arm 1 (Unasyn) or Arm 2 (ampicillin/gentamicin). She will be treated as per standard of care with tylenol, intravenous fluids, and her labor managed per physician discretion. From the time of diagnosis of chorioamnionitis until determination of treatment success or failure in the postpartum period, the patient will receive intravenous antibiotics per the protocol arm to which they have been assigned. If a patient has already been receiving ampicillin for GBS, the ampicillin will be discontinued when the study drugs are initiated. In arm 1, the study drugs will consist of Unasyn 3 grams intravenously every 6 hours, plus intravenous normal saline placebo dose every 8 hours. In arm 2, the study drugs will consist of gentamicin 1.5mg/kg intravenously every 8 hours plus ampicillin 2gm intravenously every 6 hours. For all patients, clindamycin will be given intravenously at the time of clamping of the umbilical cord in the event of a cesarean delivery, and continued as part of the antibiotic regimen as per standard of care for cesarean section in the setting of chorioamnionitis. With the exception of the saline placebo doses, both the Unasyn regimen and the ampicillin/gentamicin regimen are efficacious and widely utilized regimens for the treatment of intrapartum chorioamnionitis, and do not represent a deviation from standard of care. After delivery, if the patient experiences a treatment failure as defined below, her medical care will be managed at the discretion of the attending physician as per standard of care, and her antibiotic regimen will be unblinded. After delivery, prior to discharge from the hospital, the patient will be asked to answer a short questionnaire enquiring about side effects experienced during treatment for chorioamnionitis. The patient may receive a phone call within 14 days of delivery to assess whether she has received treatment for postpartum complications at an outside institution after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in labor or undergoing induction of labor
2. Greater than or equal to 18 years of age
3. Diagnosed with chorioamnionitis as defined by maternal temperature > or = 38.0 degrees Centigrade plus at least one of the following: maternal tachycardia (heart rate >110), fetal tachycardia (fetal heart rate baseline >160), purulent amniotic fluid, uterine tenderness.

Exclusion Criteria:

1. Allergy or adverse reaction to penicillin or ampicillin, gentamicin, or sulbactam
2. Having received antibiotics for the treatment of preterm premature rupture of membranes or other condition within the last 7 days
3. Acute or chronic renal disease or insufficiency (creatinine >1.0)
4. Hearing loss
5. Major fetal congenital anomalies or intrauterine fetal demise
6. Neutropenia
7. HIV
8. Myasthenia gravis or other neuromuscular disorder

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natali Aziz, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenberg, Mara et al. Comparison of ampicillin/sulbactam versus ampicillin/gentamicin for treatment of intrapartum chorioamnionitis: a randomized controlled trial. American Journal of Obstetrics & Gynecology , Volume 212 , Issue 1 , S145
- See also: Comparison of ampicillin/sulbactam versus ampicillin/gentamicin for treatment of intrapartum chorioamnionitis: a randomized controlled trial — http://dx.doi.org/10.1016/j.ajog.2014.10.310

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin
Started | 43 | 49
Completed | 43 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin | Total
Number analyzed (Participants) | 43 | 49 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (7.1) | 28.3 (5.6) | 28.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 49 | 92
  Male | 0 | 0 | 0
Nulliparous [Number; unit: participants] | 30 | 39 | 69
Maternal pre-existing comorbidity [Number; unit: participants] | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Defined as Resolution of Fever by 24 Hours Postpartum
Description: Proportion of patients in each arm experiencing treatment success defined as resolution of fever by 24 hours postpartum
Time Frame: Up to 24 hours after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin
Number analyzed (Participants) | 43 | 49
Participants | 43 | 49
Statistical Analysis 1: Comparison: Unasyn (Ampicillin/Sulbactam) vs Ampicillin/Gentamicin; Test type: Superiority or Other; p = 1.0, Fisher Exact

2. Secondary Outcome: Composite Maternal Morbidity
Description: Composite of maternal postpartum morbidity defined as any of the following outcomes: endometritis, clinical sepsis, pneumonia, blood transfusion or ileus.
Time Frame: Up to 6 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin
Number analyzed (Participants) | 43 | 49
Participants | 0 | 6
Statistical Analysis 1: Comparison: Ampicillin/Gentamicin; Test type: Superiority or Other; p = 0.03, Fisher Exact

3. Secondary Outcome: Neonatal Clinical Sepsis (Early Onset)
Time Frame: Up to 6 weeks after delivery
Measure: Number; unit: affected neonates
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin
Number analyzed (Participants) | 43 | 49
affected neonates | 1 | 2
Statistical Analysis 1: Comparison: Unasyn (Ampicillin/Sulbactam) vs Ampicillin/Gentamicin; Test type: Superiority or Other; p = 0.6, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 weeks after delivery.
Arm/Group | Unasyn (Ampicillin/Sulbactam) | Ampicillin/Gentamicin
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/49
Other Adverse Events (participants affected / at risk) | 2/43 | 1/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unasyn (Ampicillin/Sulbactam) (N=43) | Ampicillin/Gentamicin (N=49)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Postpartum endometritis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No